CLINICAL TRIAL: NCT03082651
Title: Investigating the Effect of Alternating Training Load and Footwear Singly or in Combination in Runners: The Alternate Run Study
Brief Title: Alternate Run Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Sports Medicine Research Foundation (Other)
Responsible Party: Principal Investigator, Jack Taunton, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H16-00858
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Overuse Injury
Keywords: Running injuries, footwear, alternating load
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Constant training/Constant footwear (Active Comparator): Group 1 - Runners will be assigned identical training sessions over a 7-day period and will perform these runs in two pairs of the same assigned neutral-cushioned running shoe (Nike Pegasus). The weekly training volume will increase on a weekly basis in order to progressively increase training load in preparation for the half-marathon event.
  Interventions: Other: Constant training; Other: Constant footwear
- Alternate training/Constant footwear (Experimental): Group 2 - Runners will perform a variation of workouts, consisting of interval/speed work, tempo runs, and long-slow distance runs throughout each 7-day period. As with Group 1, weekly training volume will increase on a weekly basis. Runners in Group 2 will perform these runs in two pairs of the same assigned neutral-cushioned running shoe (Nike Pegasus).
  Interventions: Other: Alternating run training load; Other: Constant footwear
- Constant training/Alternating footwear (Experimental): Group 3 - Runners will be assigned identical training sessions over a 7-day period but will alternate use of two different models of running shoes across successive workouts (Nike Pegasus and Nike Zoom Streak). The Zoom Streak has 10mm less midsole material, a less supportive heel counter and more flexible forefoot providing a more responsive feel to the runner.
  Interventions: Other: Alternating footwear; Other: Constant training
- Alternating training/Alternating footwear (Experimental): Group 4 - Runners will be assigned a variation of workouts throughout each 7-day period and will alternate use of two different models of running shoes across successive workouts (Nike Pegasus and Nike Zoom Streak).
  Interventions: Other: Alternating run training load; Other: Alternating footwear

INTERVENTIONS:
Other: Alternating run training load — Runners will perform a variation of workouts, consisting of interval/speed work, tempo runs, and long-slow distance runs throughout each 7-day period
  Arms: Alternate training/Constant footwear; Alternating training/Alternating footwear
Other: Alternating footwear — Runners will be assigned identical training sessions over a 7-day period but will alternate use of two different models of running shoes across successive workouts (Nike Pegasus and Nike Zoom Streak). The Zoom Streak has 10mm less midsole material, a less supportive heel counter and more flexible forefoot providing a more responsive feel to the runner.
  Arms: Alternating training/Alternating footwear; Constant training/Alternating footwear
Other: Constant training — Runners will be assigned identical training sessions over a 7-day period.
  Arms: Constant training/Alternating footwear; Constant training/Constant footwear
Other: Constant footwear — Runners perform runs in two pairs of the same assigned neutral-cushioned running shoe (Nike Pegasus).
  Arms: Alternate training/Constant footwear; Constant training/Constant footwear

SUMMARY:
The proposed study will investigate the effect of alternating footwear model and workout-type on the occurrence of running-related pain. To achieve this goal participants will be randomly assigned into one of four different groups who will perform: 1) the same workout throughout a week in the same running shoe model, 2) alternating workout-types throughout the week in the same shoe model, 3) the same workout throughout a week in alternating shoe models, and 4) alternating workouts in alternating shoes. Participants will be characterized based on body alignment, strength, injury and training history. Pain and injury status will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in this study will include adults (men and women) between the ages of 19 and 60, have been running on a regular basis (minimum once per week) over the past 6 months, are able to run for 60 minutes continuously, could tolerate 20-40km per week in training, and have not experienced a running related injury requiring a stoppage of 2-weeks or more in the past 6 months. Only neutral and pronated foot postures (Foot Posture Index between -2 and 8) will be recruited

Exclusion Criteria:

* have a history of surgery to their plantar fascia or Achilles tendon,
* have a diagnosis of osteoarthritis - or other degenerative musculoskeletal disorder - affecting the lower extremity,
* take analgesic or anti-inflammatory medication 2 or more times per week over the past 4 weeks,
* take part in high impact activities 2 or more times per week during the study period

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Running injuries | 13-weeks
  When an participant misses 3 consecutive assigned running workouts.

SECONDARY OUTCOMES:
Running-related pain | 13-weeks
  11-point numerical rating scale of overall pain associated with running
Region specific running-related pain | 13-weeks
  Numerical rating scale for pain at selected anatomical locations: gluteal, low back, groin, thigh, hamstring, knee, calf, Achilles, ankle, foot.
Footwear comfort | 13-weeks
  11-point rating of footwear comfort
Run Quality | 13-weeks
  Study specific 11-point measure of how the footwear used affected each run's quality

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Sports Medicine, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No